CLINICAL TRIAL: NCT03154398
Title: Thyroid Dysfunction in Patients With Type 2 Diabetes With Early Diabetic Nephropathy.
Acronym: AssuitU
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, maria hamdy, principal investigator, Assiut University
Other Study IDs: Assiut1991
Record Dates: First submitted 2017-05-14; First posted 2017-05-16 (Actual); Last update posted 2021-02-15 (Actual); Status verified 2021-02

CONDITIONS: Evaluation Thyroid Functions in Diabetic Patient
Keywords: evaluation of thyroid function in diabetes patients

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1: case control

SUMMARY:
Diabetes Mellitus is the most common disorder seen. The impact of this disease on the quality of life, and on morbidity and mortality through the complications that affect the small and large vessels resulting in retinopathy, nephropathy, neuropathy, and ischemic heart disease has been emphasized by the findings of the national commission (USA) on diabetes .

So, there was curiosity to understand and learn the association of this disorder with another common endocrine gland function that is thyroid gland . The association between these two disorders has long been recognized although the prevalence of thyroid dysfunction in diabetic population varies widely between studies. With insulin and thyroid hormone being intimately involved in cellular metabolism and thus excess or deficit of these hormones result in functional derangement of the other .

Diabetic patients have higher prevalence of thyroid disorder when compared with the normal population. Diabetic women are more frequently affected than men and hypothyroidism is more common than thyrotoxicosis.

As Hyperthyroidism impairs glycemic control in diabetic subjects, while hypothyroidism may increase susceptibility to hypoglycemia thus complicating diabetes management so Severe diabetic complications where noted in patients with sub- clinical hypothyroidism . Sub-clinical hypothyroidism is an independent risk factor for development of diabetic nephropathy.

DETAILED DESCRIPTION:
Recognition and treatment of thyroid dysfunction in diabetic patients will benefit glycemic control and improve general well-being Diabetic nephropathy, a major microvascular complication of type 2 diabetes mellitus, is an important cause of chronic kidney disease. It results from interactions between hemodynamic and metabolic factors.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes mellitus and with diabetic nephropathy.

Exclusion Criteria:

* 1) Insulin dependent diabetes 2) Patients with:

  * Gestational diabetes mellitus.
  * Steroid induced Diabetes.

    3) Thyroid disease

Ages: 40 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: type 2 diabetes with early nephropthy
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2019-05-01 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
the percentage of patients progress to advanced diabetic nephropathy | one year

CONTACTS AND LOCATIONS:
Overall Officials: maria hamdy, Study Director — Assiut University
Locations (1):
- Assuit University, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No
evaluate thyroid dysfunction in patients with diabetes in diabetic nephropathy